CLINICAL TRIAL: NCT00954512
Title: A Dose-Escalation Study to Evaluate the Safety and Tolerability of SCH 717454 in Combination With Different Treatment Regimens in Subjects With Advanced Solid Tumors (Phase 1B/2; Protocol No. P04722)
Brief Title: Study of Robatumumab (SCH 717454, MK-7454) in Combination With Different Treatment Regimens in Participants With Advanced Solid Tumors (P04722, MK-7454-004)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04722; MK-7454-004 (Other: Merck Protocol Number); 2009-011101-16 (EudraCT Number)
Record Dates: First submitted 2009-07-23; First posted 2009-08-07 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms
Keywords: Antibodies, neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin; Epirubicin; Trastuzumab; Everolimus; Gemcitabine; robatumumab; Cetuximab; Paclitaxel; Cisplatin; Fluorouracil; Erlotinib Hydrochloride; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Regimen A: FOLFIRI (± Cetuximab) + Robatumumab (Experimental): Participants with colorectal adenocarcinoma receive FOLFIRI (Irinotecan 180 mg/m^2+ folinic acid 400 mg/m^2+ 5-fluorouracil [5-FU] 400 mg/m^2 bolus followed by 2400 mg/m^2 intravenous [IV] infusion over 46 hours) (± cetuximab initial dose of 400 mg/m^2 IV followed by once-weekly doses of 250 mg/m^2 IV) PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 2-week cycle.
  Interventions: Biological: Robatumumab; Biological: Cetuximab; Drug: 5-FU; Drug: Irinotecan; Drug: Folinic Acid
- Regimen B: Carboplatin + Paclitaxel + Robatumumab (Experimental): Participants with non-small cell lung cancer receive carboplatin administered at an area under the curve (AUC) of 6 mg/mL/min IV PLUS paclitaxel 225 mg/m^2 IV PLUS robatumumab 15 mg/kg IV on Day 1 of each 3-week cycle.
  Interventions: Drug: Carboplatin; Biological: Robatumumab; Drug: Paclitaxel
- Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab (Experimental): Participants with gastric adenocarcinoma receive epirubicin 50 mg/m^2 IV PLUS cisplatin 60 mg/m^2 IV PLUS 5-FU 200 mg/m^2/day administered via a 21-week continuous IV infusion PLUS robatumumab 15 mg/kg IV on Day 1 of each 3-week cycle.
  Interventions: Drug: Epirubicin; Biological: Robatumumab; Drug: Cisplatin; Drug: 5-FU
- Regimen D: Trastuzumab + Robatumumab (Experimental): Participants with human epidermal growth factor receptor 2 positive (Her2+) breast cancer receive trastuzumab 4 mg/kg IV once every week PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 4-week cycle.
  Interventions: Biological: Trastuzumab; Biological: Robatumumab
- Regimen E: mTor Inhibitor (Everolimus) + Robatumumab (Experimental): Participants with renal cell cancer receive mammalian target of rapamycin (mTor) inhibitor (everolimus) 10 mg orally once per day PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 4-week cycle.
  Interventions: Drug: Everolimus; Biological: Robatumumab
- Regimen F: Gemcitabine (± Erlotinib) + Robatumumab (Experimental): Participants with pancreatic adenocarcinoma receive gemcitabine 1000 mg/m^2 IV on Days 1, 8, 15, 22, 29, 36, and 43 in Cycle 1 and on Days 1, 8 and 15 in subsequent cycles (± erlotinib 100 mg per day orally) PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 4-week cycle. (Cycle 1 is 8 weeks.)
  Interventions: Drug: Gemcitabine; Biological: Robatumumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Carboplatin
  Arms: Regimen B: Carboplatin + Paclitaxel + Robatumumab
Drug: Epirubicin
  Arms: Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab
Biological: Trastuzumab
  Arms: Regimen D: Trastuzumab + Robatumumab
Drug: Everolimus
  Arms: Regimen E: mTor Inhibitor (Everolimus) + Robatumumab
Drug: Gemcitabine
  Arms: Regimen F: Gemcitabine (± Erlotinib) + Robatumumab
Biological: Robatumumab — In Part 1, robatumumab was to be administered at 10 mg/kg, 15 mg/kg (for Regimens B and C), or 20 mg/kg together with the assigned standard treatment. For Part 2, robatumumab was to be administered at the dose selected during Part 1, based upon the maximum tolerated dose (MTD) or maximum administered dose (MAD), pharmacokinetic (PK) and pharmacodynamic (PD) data.
Biological: Cetuximab
  Arms: Regimen A: FOLFIRI (± Cetuximab) + Robatumumab
Drug: Paclitaxel
  Arms: Regimen B: Carboplatin + Paclitaxel + Robatumumab
Drug: Cisplatin
  Arms: Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab
Drug: 5-FU
  Arms: Regimen A: FOLFIRI (± Cetuximab) + Robatumumab; Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab
Drug: Erlotinib
  Arms: Regimen F: Gemcitabine (± Erlotinib) + Robatumumab
Drug: Irinotecan
  Arms: Regimen A: FOLFIRI (± Cetuximab) + Robatumumab
Drug: Folinic Acid
  Arms: Regimen A: FOLFIRI (± Cetuximab) + Robatumumab

SUMMARY:
This is a Phase 1B/2, non-randomized, dose-escalation, multicenter, open-label study designed to evaluate the safety and tolerability of robatumumab (SCH 717454, MK-7454) in combination with standard treatment in participants with advanced solid tumors to be conducted in conformance with Good Clinical Practices.

Six different treatment regimens will be investigated in combination with robatumumab.

The study will be divided into two parts. Part 1 will consist of initial safety evaluation and dose-finding of robatumumab in combination with each treatment regimen. Part 2 will consist of an expansion of each robatumumab regimen at a newly established dose level, to better define safety, tolerability, and initial efficacy in specific target populations.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the study.
* Be ±18 years of age of either sex and of any race/ethnicity;
* Part 1: Have a histologically or cytologically confirmed advanced malignant solid tumor;
* Part 2: Have a histologically or cytologically confirmed, with measurable disease (as defined by Response Evaluation Criteria in Solid Tumors [RECIST]), advanced, malignant solid tumor.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of <=2.
* Have adequate organ function within 3 weeks prior to first study drug administration.

Exclusion Criteria:

* Not have known treated or untreated leptomeningeal metastasis or a metastatic central nervous system lesion.
* Not have a history of another malignancy
* Not have received prior therapy with any anti-insulin-like growth factor receptor 1 (anti-IGF-1R) monoclonal antibody.
* Not have received radiation therapy within 2 weeks prior to first study drug administration.
* Not have received radiation therapy to >25% of his/her total bone marrow during his/her lifetime.
* Not have undergone major surgery within 3 weeks prior to first study drug administration.
* Not have known human immunodeficiency virus (HIV) infection or a known HIV-related malignancy.
* Not have known active hepatitis B or C.
* Not have any serious or uncontrolled infection.
* Not have uncontrolled diabetes mellitus.
* Not have had any of the following within 6 months prior to first study drug administration: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality, cerebrovascular accident or transient ischemic attack, or seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2011-06-07 (Actual); Study Completion 2011-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synospsi Links — http://www.merck.com/clinical-trials/study.html?id=P04722&kw=P04722&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: FOLFIRI (± Cetuximab) + Robatumumab: Participants with colorectal adenocarcinoma receive FOLFIRI (Irinotecan 180 mg/m^2+ folinic acid 400 mg/m^2+ 5-FU 400 mg/m^2 bolus followed by 2400 mg/m^2 IV infusion over 46 hours) (± cetuximab initial dose of 400 mg/m^2 IV followed by once-weekly doses of 250 mg/m^2 IV) PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 2-week cycle.
- Regimen B: Carboplatin + Paclitaxel + Robatumumab: Participants with non-small cell lung cancer receive carboplatin administered at an AUC of 6 mg/mL/min IV PLUS paclitaxel 225 mg/m^2 IV PLUS robatumumab 15 mg/kg IV on Day 1 of each 3-week cycle.
- Regimen D: Trastuzumab + Robatumumab: Participants with Her2+ breast cancer receive trastuzumab 4 mg/kg IV once every week PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 4-week cycle.
- Regimen E: mTor Inhibitor (Everolimus) + Robatumumab: Participants with renal cell cancer receive mTor inhibitor (everolimus) 10 mg orally once per day PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 4-week cycle.
Period: Overall Study
Arm/Group | Regimen A: FOLFIRI (± Cetuximab) + Robatumumab | Regimen B: Carboplatin + Paclitaxel + Robatumumab | Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab | Regimen D: Trastuzumab + Robatumumab | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab | Regimen F: Gemcitabine (± Erlotinib) + Robatumumab
Started | 2 | 3 | 0 | 2 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 0 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Progression of Disease | 2 | 1 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A: FOLFIRI (± Cetuximab) + Robatumumab | Regimen B: Carboplatin + Paclitaxel + Robatumumab | Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab | Regimen D: Trastuzumab + Robatumumab | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab | Regimen F: Gemcitabine (± Erlotinib) + Robatumumab | Total
Number analyzed (Participants) | 2 | 3 | 0 | 2 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (2.8) | 54.0 (4.4) |  | 48.0 (2.8) | 53.3 (13.5) | 70.8 (3.0) | 56.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 |  | 2 | 1 | 3 | 11
  Male | 0 | 0 |  | 0 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Number of Participants With Each Type of Response Evaluation Criteria in Solid Tumors (RECIST)-Determined Overall Best Response
Description: Overall best response was determined by RECIST criteria. Types of overall response could be: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Assessable (NA) or Incomplete Response/Stable Disease (IR/SD).
Time Frame: Up to ~30 days after the final dose of robatumumab (Up to ~14 months)
Population: The All Treated Set (efficacy) consisted of all participants who received ≥1 dose of study drug and were evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Regimen A: FOLFIRI (± Cetuximab) + Robatumumab | Regimen B: Carboplatin + Paclitaxel + Robatumumab | Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab | Regimen D: Trastuzumab + Robatumumab | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab | Regimen F: Gemcitabine (± Erlotinib) + Robatumumab
Number analyzed (Participants) | 2 | 3 | 0 | 2 | 3 | 2
Participants
  Complete Response (CR) | 0 | 0 |  | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 |  | 0 | 0 | 0
  Stable Disease (SD) | 0 | 2 |  | 1 | 2 | 1
  Progressive Disease (PD) | 2 | 1 |  | 1 | 1 | 1
  Not Assessable (NA) | 0 | 0 |  | 0 | 0 | 0
  Incomplete Response/Stable Disease (IR/SD) | 0 | 0 |  | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to this study drug. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to ~30 days after the final dose of robatumumab (Up to ~14 months)
Population: The All Treated Set (safety) consisted of all participants who received ≥1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Regimen A: FOLFIRI (± Cetuximab) + Robatumumab | Regimen B: Carboplatin + Paclitaxel + Robatumumab | Regimen C: Epirubicin + Cisplatin + 5-FU + Robatumumab | Regimen D: Trastuzumab + Robatumumab | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab | Regimen F: Gemcitabine (± Erlotinib) + Robatumumab
Number analyzed (Participants) | 2 | 3 | 0 | 2 | 4 | 4
Participants | 2 | 3 |  | 2 | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to ~30 days after the final dose of robatumumab (Up to ~14 months)
Description: The All Treated Set consisted of all participants who received ≥1 dose of study drug.
Groups:
- Regimen A: FOLFIRI (+/- Cetuximab) + Robatumumab: Participants with colorectal adenocarcinoma receive FOLFIRI (Irinotecan 180 mg/m^2+ folinic acid 400 mg/m^2+ 5-FU 400 mg/m^2 bolus followed by 2400 mg/m^2 IV infusion over 46 hours) (± cetuximab initial dose of 400 mg/m^2 followed by once-weekly doses of 250 mg/m^2) PLUS robatumumab 10 mg/kg or 20 mg/kg IV. Each cycle is 2 weeks.
- Regimen F: Gemcitabine (+/- Erlotinib) + Robatumumab: Participants with pancreatic adenocarcinoma receive gemcitabine 1000 mg/m^2 on Days 1, 8, 15, 22, 29, 36, and 43 (± erlotinib 100 mg per day) PLUS robatumumab 10 mg/kg or 20 mg/kg IV. Each cycle is 8 weeks.
Arm/Group | Regimen A: FOLFIRI (+/- Cetuximab) + Robatumumab | Regimen B: Carboplatin + Paclitaxel + Robatumumab | Regimen D: Trastuzumab + Robatumumab | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab | Regimen F: Gemcitabine (+/- Erlotinib) + Robatumumab
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/3 | 1/2 | 2/4 | 2/4
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 2/2 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: FOLFIRI (+/- Cetuximab) + Robatumumab (N=2) | Regimen B: Carboplatin + Paclitaxel + Robatumumab (N=3) | Regimen D: Trastuzumab + Robatumumab (N=2) | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab (N=4) | Regimen F: Gemcitabine (+/- Erlotinib) + Robatumumab (N=4)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: FOLFIRI (+/- Cetuximab) + Robatumumab (N=2) | Regimen B: Carboplatin + Paclitaxel + Robatumumab (N=3) | Regimen D: Trastuzumab + Robatumumab (N=2) | Regimen E: mTor Inhibitor (Everolimus) + Robatumumab (N=4) | Regimen F: Gemcitabine (+/- Erlotinib) + Robatumumab (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (11) | 3 (12)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (10)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 3 (4)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
GINGIVITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (4) | 0 (0) | 3 (3) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (9)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (4) | 3 (9) | 1 (2) | 1 (1) | 1 (2)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
HYPERPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (9) | 2 (2) | 2 (3) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 1 (2) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
PHANTOM PAIN (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANTICIPATORY ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL BLISTERING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.